CLINICAL TRIAL: NCT06927804
Title: Utilization of Virtual Reality to Support Patient Comfort and Reduce Stress During the Implantation of a Subcutaneous Venous Port Prior to the Initiation of Oncological Treatment
Brief Title: Utilization of Virtual Reality to Increase Comfort and Reduce Procedural Distress During Port Insertion Into the Body
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FNO-ONK-VIREPO; LERCO Research Project (Other: University Hospital Ostrava)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Oncology Patients
Keywords: Virtual reality; subcutaneous venous port; anxiety; stress; pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This interventional study compares two approaches to subcutaneous venous port implantation in adult oncology patients: standard care versus standard care with the use of immersive virtual reality to reduce pain, stress, and anxiety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): In patients randomized in this study arm, a virtual reality device will be used during the subcutaneous port implantation procedure.
  Interventions: Procedure: Virtual reality intervention
- Non-VR Group (Active Comparator): In patients randomized in this study arm, no virtual reality device will be used during the subcutaneous port implantation procedure.
  Interventions: Procedure: Standard Care (in control arm)

INTERVENTIONS:
Procedure: Virtual reality intervention — A virtual reality device will be used in one study arm during the implantation of the subcutaneous port.
  Arms: VR Group
Procedure: Standard Care (in control arm) — Patients in this study arm will receive standard care, without the use of VR.
  Arms: Non-VR Group

SUMMARY:
This randomised controlled study evaluates whether virtual reality (VR) can support patient comfort and help reduce anxiety and stress during subcutaneous venous port implantation in adult oncology patients. Patients will be assigned to standard care or standard care with VR intervention.

Subjective and objective measures of stress and discomfort will be collected, including the Visual Analog Scale (VAS) for self-reported procedural discomfort, physiological parameters (blood pressure, heart rate, variability), the STAI-6 questionnaire, and salivary cortisol.

The study aims to explore the potential of VR as a non-pharmacological, immersive tool to improve procedural experience and reduce psychological distress in patients undergo-ing minor oncological procedures.

DETAILED DESCRIPTION:
The implantation of a subcutaneous venous port is a minor surgical procedure that has become a routine component of oncological care. It is indicated in cases where the expected duration of systemic treatment exceeds six months and where there is a significant risk of damage to the peripheral venous system due to chemotherapy.

Although generally well tolerated, the procedure is invasive and often associated with varying degrees of psychological stress, discomfort, and procedural anxiety. It is performed under local anaesthesia, often accompanied by mild sedation, and typically lasts about 60 minutes.

The application of virtual reality (VR) during such procedures represents a non-pharmacological approach that may help mitigate psychological stress and procedural discomfort by immersing the patient in a calming, engaging virtual environment. VR-based distraction techniques have previously been shown to promote relaxation and improve perceived comfort in various clinical settings.

The aim of this randomised study is to assess the impact of immersive VR on patient comfort, anxiety, and stress during venous port implantation in adult oncology patients.

Two study arms will be compared:

* control group (standard care with local anaesthesia and optional symptomatic sedation)
* VR group (standard care with the addition of immersive VR during the procedure)

Discomfort Assessment: Procedural discomfort will be evaluated using the Visual Analog Scale (VAS), administered in a standardised three-point timeline:

* 30 minutes before the procedure
* during the procedure (at a predefined time point)
* 30 minutes after the procedure

Physiological indicators associated with stress and procedural discomfort will also be recorded at these same time points:

* blood pressure
* heart rate
* heart rate variability

Measurements will follow standardized protocols and consistent conditions.

Anxiety and Stress Evaluation: Psychological stress and anxiety will be assessed using both subjective and objective measures:

* STAI-6 questionnaire administered 30 minutes before and after the procedure
* Salivary cortisol collected before the procedure (baseline), midway through, and 30 minutes after

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Signed Informed Consent Form
* Patients Indicated for oncology treatment administration using subcutaneous port

Exclusion Criteria:

* Not signing of the Informed Consent Form
* Patients < 18 years of age
* Patients unsuitable for subcutaneous port implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the level of pain | 2 hours
  Changes in the level of pain in patients undergoing sub-cutaneous venous port implantation will be measured using the Visual Analog Scale (VAS). The assessment will be performed at three standardized time points: 30 minutes before, during, and 30 minutes after the procedure.
Changes in the level of stress and anxiety | 2 hours
  Changes in the level of stress and anxiety in patients undergoing sub-cutaneous venous port implantation will be measured using the State-Traint Anxiety Inventory (STAI-6) questionnaire. The assessment will be performed at three standardized time points: 30 minutes before, during, and 30 minutes after the procedure.
Changes in the level of procedural discomfort | 2 hours
  Subjective discomfort will be measured using the Visual Analog Scale (VAS) at three standardised time points. The scale is a straight, 10-centimetre line with descriptive anchors at each end, like "no pain" and "worst pain imaginable".

SECONDARY OUTCOMES:
Changes in blood pressure | 2 hours
  Changes in blood pressure in patients undergoing sub-cutaneous venous port implantation will be observed at three standardized time points: 30 minutes before, during, and 30 minutes after the procedure and measured in mmHg.
Changes in heart rate | 2 hours
  Changes in heart rate in patients undergoing sub-cutaneous venous port implantation will be observed at three standardized time points: 30 minutes before, during, and 30 minutes after the procedure and measured in beats per minute.
Changes in heart rate variability | 2 hours
  Changes in heart rate variability in patients undergoing sub-cutaneous venous port implantation will be observed at three standardized time points: 30 minutes before, during, and 30 minutes after the procedure and measured in beat-to-beat intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Lukáš Knybel, Ing., PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Gokce E, Arslan S. Effects of virtual reality and acupressure interventions on pain, anxiety, vital signs and comfort in catheter extraction processes for patients undergoing coronary angiography: A randomized controlled trial. Int J Nurs Pract. 2023 Dec;29(6):e13176. doi: 10.1111/ijn.13176. Epub 2023 Jul 4. PMID 37403339
- [Background] Menekli T, Yaprak B, Dogan R. The Effect of Virtual Reality Distraction Intervention on Pain, Anxiety, and Vital Signs of Oncology Patients Undergoing Port Catheter Implantation: A Randomized Controlled Study. Pain Manag Nurs. 2022 Oct;23(5):585-590. doi: 10.1016/j.pmn.2022.03.004. Epub 2022 Mar 31. PMID 35367144